CLINICAL TRIAL: NCT02899806
Title: Impact of a Video Explaining Epidural Analgesia in Obstetrics in Terms of Satisfaction, Understanding and Anxiety: A Prospective Randomised Trial
Brief Title: Impact of a Video Explaining Epidural Analgesia in Obstetrics
Acronym: VIDEOCLIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Principal Investigator, Marion ANDREOLETTI, Physician, Centre Hospitalier Intercommunal Creteil
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: VIDEOCLIP
Record Dates: First submitted 2016-08-30; First posted 2016-09-14 (Estimated); Last update posted 2020-07-16 (Actual); Status verified 2017-07

CONDITIONS: Difficulty Processing Information
Keywords: Video Information; Satisfaction; Anxiety; Epidural Analgesia; Comprehension; delivery
MeSH Terms: conditions — Personal Satisfaction; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paper (Placebo Comparator): Information about epidural analgesia by oral and paper sheep given by anesthesist in programed consultation
  Interventions: Other: Written Information
- Video (Experimental): Video information in addition to oral and written information gave by anesthesist in programed consultation
  Interventions: Other: Written Information; Other: Video Information

INTERVENTIONS:
Other: Written Information — A written information on peridural anesthesia is delivered
Other: Video Information — A link to a video explaining peridural anesthesia is delivered to the pregnant woman. The patient can watch the video several times.
  Arms: Video

SUMMARY:
The aim of this study was to investigate the impact of multimedia information on epidural anesthesia. Pregnant women were randomly assessed to get a video information in addition to an oral and written information on epidural anesthesia. Maternal satisfaction concerning the quality of the information as well their anxiety and understanding of the procedure were assessed and compared in both groups.

DETAILED DESCRIPTION:
The information in anesthesia consultation is mandatory. Few studies have investigated the impact of multimedia preoperative information in terms of satisfaction, comprehension and anxiety, with conflicting results. None have evaluated the contribution of a video explaining epidural analgesia in obstetrics. This study compared two types of information given in anesthesia consultation: an oral and written information (group P) versus oral, written and video information (group V). The main objective was maternal satisfaction, the secondary objectives were understanding and anxiety.

This is a common care, prospective and randomized study, conducted between September 2015 and February 2016 in the Creteil Intercommunal Hospital Center (CHIC) and accepted by the ethics committee Paris V. After information, not opposition of women who accepted to participated was collected. Oral information on epidural analgesia was provided in consultation by the anesthesiologist, with delivery of a written information sheet. The video made at CHIC in 2015, was transmitted, in addition, by email to patients randomized in the group V for she could look it at their convenience. Satisfaction and anxiety were evaluated by numerical scale from 0 to 10 and comprehension by multiple choice questions with a final score of 10. These three criteria were also evaluated in an emergency context in which women received oral and written information (group U). Evaluation questionnaires were given during the anesthesia consultation and recovered during the hospitalization after childbirth.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman
* Affiliated to social security system
* Understanding French language
* Internet access
* >18 years old and not subject to a measure of legal protection

Exclusion Criteria:

* Contre indications to epidural
* Refusal to participate in the study
* Not affiliated with the Social Security system
* No understanding French
* No access to Internet
* Patient minor or under legal protection

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 301 (Actual)
Dates: Start 2015-09; Primary Completion 2015-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Satisfaction evaluated by numerical scale from 0 to 10 | during the 48 hour after delivery

SECONDARY OUTCOMES:
Comprehension was evaluated by by multiple choice questions with a final score of 10 | during the 48 hour after delivery
Anxiety was evaluated by numerical scale from 0 to 10 | during the 48 hour after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Marion ANDREOLETTI, MD, Principal Investigator — CHI de Créteil
Locations (1):
- Centre Hospitalier Intercommunal, Créteil, France

IPD SHARING:
Plan to Share IPD: No